CLINICAL TRIAL: NCT03587337
Title: Risk of Microbial Translocation in Patients Undergoing Per-Oral Endoscopic Myotomy (POEM) for Achalasia: Antibiotic Prophylaxis or Short-therapy
Acronym: POEM-MT01
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1789
Record Dates: First submitted 2018-02-19; First posted 2018-07-16 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-07

CONDITIONS: Achalasia
Keywords: Per-Oral Endoscopy Myotomy; Microbial Translocation
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylaxis
  Interventions: Other: POEM
- Antibiotic tp
  Interventions: Other: POEM

INTERVENTIONS:
Other: POEM — Pt. are going to submit a POEM procedure.

SUMMARY:
Background: Achalasia is a primary rare esophageal motor disorder of the esophagus (annual incidence of 1:100,000 persons). Recently, a new endoscopic technique, Per-Oral Endoscopic Myotomy (POEM), has been introduced with excellent success rates. Several studies have evaluated complications of POEM but there is a lack of knowledge on the potential risk of bacteremia or microbial translocation during the endoscopic intervention and, also, there aren't evidences regarding the use of antibiotics before/after POEM. Microbial translocation (MT) is the passage of both viable and nonviable microbes across the anatomically intact GI barrier to the mesenteric lymph nodes, and possibly other tissues. Gram-negative bacteria contain lipopolysaccharides (LPSs) coating their thin peptidoglycan cell wall. The presence of LPS, an endotoxin, in the plasma has been correlated to sepsis and septic shock through the activation of the inflammatory host defence via binding to soluble CD14 (sCD14) which initiates downstream cytokines (like IL-6, IL-8 and tumor necrosis factor (TNF-α)) and, also, through the production of sCD14 and LPS-binding protein (LBP) by the innate immune system.

Objectives: Considering POEM a clean-contaminated procedure, it should be assessed whether the post-POEM fever or systemic inflammation is a cytokinin-mediated or an infection-related fever. Thus, aim of the study is to evaluate the presence of inflammation mediators, bacteremia and microbial translocation post POEM, to guide future antibiotic prophylaxis/therapy in patients undergoing this procedure.

Methods: All patients who will undergo POEM at _Investigator's Department from June 2017 to June 2019 will be enrolled in a prospective, interventional randomized clinical trial (RCT). Patients will be randomized in two groups. The Group A, prophylaxis group, will receive antibiotics (Cefazolin 2 gr i.v.) only before procedure whereas Group B, short therapy group, will receive antibiotics before POEM (Cefazolin 2 gr i.v.), continued for the first 24 hours and then per os (Amoxicilline/Clavulanic Acid 3 gr/die) for 3 days. For each patient we will be evaluated: dosage of IL-6, IL-1β, TNF-α, sCD4, LPB, LPS and blood cultures.

Expected results: we expect that the prophylaxis group vs short therapy group, has a prevalence of fever and/or systemic inflammation not higher than 10% difference of the fever related to the procedure.

ELIGIBILITY:
Inclusion criteria:

* patients with had a diagnosis of achalasia defined by symptoms,HR manometry and X-ray accordingly to guidelines,who have no absolute contraindications to undergo interventions under general anesthesia
* age over 18 years old
* ability to provide and to give informed consent
* body temperature under 37°C on the day before and just before POEM

Exclusion criteria:

* antibiotic use within 1 week before the procedure
* patients who had chronic inflammatory diseases (such as rheumatic arthritis or inflammatory bowel diseseas) and/or known neoplasia
* inability to obtain written informed consent
* patient unwilling to take part in the study
* impossibility to be subjected to the invasive endoscopic procedure or general anesthesia for the presence of comorbidities
* known allergy to drugs provided in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: patients older than 18, with esophageal achalasia (diagnosed accordingly to the international guidelines) scheduled for POEM, who are willing to participate in a RCT and who are able able to give informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Presence of inflammation mediators, bacteremia and micro translocation | 18 Months
  Assesment of fever (TC>38°C) and systemic inflammation (increased in white blood cells (WBC) and/or protein C-reactive (PCR)) that may occur following POEM

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maselli R, Oliva A, Badalamenti M, Galtieri PA, Belletrutti PJ, Spadaccini M, Nicoletti R, Finati E, Vetrano S, Fosso F, Correale C, Pellegatta G, Hassan C, Repici A. Single-dose versus short-course prophylactic antibiotics for peroral endoscopic myotomy: a randomized controlled trial. Gastrointest Endosc. 2021 Nov;94(5):922-929. doi: 10.1016/j.gie.2021.05.045. Epub 2021 Jun 11. PMID 34119499

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03587337/Prot_SAP_000.pdf